CLINICAL TRIAL: NCT00001136
Title: A Multi-Centered Phase 1 Trial to Evaluate the Memory Responses to a Single Boosting Vaccination With ALVAC-HIV vCP205 in Volunteers Who Have Previously Received Poxvirus-Based Vaccines
Brief Title: A Study of the Effectiveness of an HIV Vaccine (ALVAC vCP205) to Boost Immune Functions in HIV-Negative Volunteers Who Have Already Received an HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: AVEG 038; 10586 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2000-01-25; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Injections, Intramuscular; HIV-1; AIDS Vaccines; CD4-Positive T-Lymphocytes; CD8-Positive T-Lymphocytes; T-Lymphocytes, Cytotoxic; Gene Products, gag; HIV Seronegativity; Immunologic Memory; Antibodies, Viral; Genetic Vectors; Gene Products, env; Poxviridae; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC-HIV MN120TMG (vCP205)

SUMMARY:
The purpose of this study is to see if it is safe to give an HIV vaccine (vCP205) to volunteers who received an HIV vaccine at least 2 years ago, and to study how the immune system responds to this vaccine.

Vaccines are given to people to try to resist infection or prevent disease. There are a number of different HIV vaccines that are currently being tested. The vaccines that seem to be the most promising are canarypox vaccines, known as ALVAC vaccines; the vaccine tested in this study is ALVAC-HIV vCP205. This study will look at the safety of the vaccine and how the immune system responds to it.

DETAILED DESCRIPTION:
Vaccines may provide a route of therapy against HIV-1 infections by boosting the immune system responses. An artificially constructed HIV-1 vaccine (NYCBH), using vaccinia virus as its vector, has the advantage of conferring both cellular and humoral immune responses that are long-lived. Studies have shown that a second artificially constructed vector vaccine, HIV-1 canarypox (vCP205), also increases CD8+ cytotoxic T lymphocyte (CTL) activity, a cell-mediated immune response. Yet, immune responses are not boosted in volunteers previously vaccinated with vaccinia-based HIV-1 vaccines when a second vaccination with the same vaccine is given. One theory for vaccinia vaccine's failure is that immunologic barriers by antibodies to the vector itself may be responsible. This study examines the effectiveness of boosting the immune responses following vCP205 vaccination in the following: 1) volunteers who were previously immunized with vCP205 vaccine who may or may not have shown increased immune responses following the first immunization, and 2) volunteers who were previously immunized with NYCBH vaccine.

Upon study entry volunteers receive one injection of ALVAC-HIV vCP205. Temperature and symptoms should be recorded by the volunteer each day for 2 days and reported to the clinic staff. Volunteers will have seven clinic visits for drawing blood, collecting urine specimens, and performing clinical evaluations. At Month 3 HIV testing will be done. Volunteers will be followed for 3 months, with a passive follow-up call at the end of a year and once or twice a year for the next 5 years. Counseling on avoidance of HIV infection and pregnancy will be done.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are 18-60 years old.
* Are willing to use adequate birth control for 1 month before study entry and during the study.
* Have a CD4 count of at least 400 cells/mm3.
* Have a normal medical history and physical examination.
* Are available for 3 months of follow-up.
* Have participated in AVEG Protocol 014C or 022A and received all the scheduled vaccinations 24 or more months before this study, or have never participated in HIV-vaccine studies.
* Are HIV-negative within 8 weeks of study entry.
* Are negative for hepatitis B surface antigen.

Exclusion Criteria

You will not be eligible for this study if you:

* Are pregnant or breast-feeding.
* Have a history of an immune system problem, any long-term illness, or any autoimmune disease.
* Have a history of using medications which affect your immune system.
* Have a history of cancer, except if it has been removed with surgery and cure is most likely.
* Have a medical or mental condition which interferes with the study.
* Have a job or work which interferes with the study.
* Have ever attempted suicide, thought of attempting suicide, or have a severe mental condition.
* Have received vaccines within 60 days of study entry.
* Have used experimental drugs within 30 days prior to study entry.
* Have received any blood products, such as immunoglobulin, in the last 6 months.
* Have active syphilis.
* Have active tuberculosis.
* Have any history of severe allergic reactions, including reactions to vaccines.
* Have an allergy to egg products or neomycin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Evans, Study Chair
Locations (6):
- United States (6):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington